CLINICAL TRIAL: NCT06091891
Title: Effect of ROTEM®-Guided Algorithm for Tranexamic Acid Administration in Pediatric Scoliosis Surgery: a Prospective Randomized Controlled Trial
Brief Title: Tranexamic Acid in Pediatric Scoliosis Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Eun-hee Kim, clinical associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2308-113-1459
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Scoliosis
MeSH Terms: conditions — Scoliosis | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Drug: Tranexamic acid
- ROTEM-guided (Experimental)
  Interventions: Drug: Tranexamic acid infusion under ROTEM-guidance

INTERVENTIONS:
Drug: Tranexamic acid — Without ROTEM-guidance, we maintain tranexamic acid infusion at 10mg/kg/h until the end of the surgery.
  Arms: Control
Drug: Tranexamic acid infusion under ROTEM-guidance — If diffuse bleeding occurs during surgery, we perform ROTEM testing and administer tranexamic acid based on the test results.
  Arms: ROTEM-guided

SUMMARY:
This study aims to investigate whether intraoperative administration of tranexamic acid based on ROTEM® (Rotational Thromboelastometry), in pediatric patients undergoing scoliosis surgery, results in a difference in intraoperative blood loss when compared to the prophylactic administration of tranexamic acid.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing scoliosis surgery under the age of 18

Exclusion Criteria:

* Patients with coagulation disorders
* Patients at an increased risk of thrombosis
* Patients with a history of epilepsy or brain surgery
* Patients with a previous allergic reaction or anaphylaxis history to tranexamic acid
* Severe liver or kidney impairment
* Other cases deemed inappropriate by the researcher

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-10-16 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
intraoperative bleeding loss | during surgery (From induction of anesthesia to when the patient leaves the operating room.)
  total volume of blood loss during surgery determined by anesthesiologist

SECONDARY OUTCOMES:
RBC blood transfusion | during surgery (From induction of anesthesia to when the patient leaves the operating room.)
  intraoperative red blood cell volume of transfused during surgery per hour
urine output | during surgery (From induction of anesthesia to when the patient leaves the operating room.)
  intraoperative total urine output during surgery per hour
Other blood transfusion | during surgery (From induction of anesthesia to when the patient leaves the operating room.)
  Volume of blood cells transfused during surgery per hour, such as FFP, platelets, and cryoprecipitates.
postoperative viscoelastic whole blood profile | 1 hours from the end of surgery
  CT, CFT, A10, MCF, ML in EXTEM and CT, CFT, A10, MCF, ML in FIBTEM at the end of surgery
JP drain | 24 hours from the end of surgery
  total JP drain for 24 hours after the end of surgery
IL-6 | 1 hours from the end of surgery
  the change in IL-6 values before and after surgery
total tranexamic acid dose | during surgery (From induction of anesthesia to when the patient leaves the operating room.)
  Total amount of tranexamic acid used during surgery
postoperative complications | 2 weeks from the end of surgery
  Presence of unexpected ICU admissions, mechanical ventilation, respiratory complications, convulsions, and thromboembolic events.

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Bin Park, Study Director — Seoul National University Hospital
Locations (1):
- Seoul national university hospital, Seoul, South Korea